CLINICAL TRIAL: NCT04892784
Title: THE EFFECT OF PRESS TACK NEEDLE ACUPUNCTURE ON THE REDUCTION OF POST-EXERCISE BLOOD LACTIC ACID LEVELS IN SPORT STUDENTS
Brief Title: THE EFFECT OF ACUPUNCTURE ON THE BLOOD LACTIC ACID LEVELS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Wahyuningsih Djaali, Student, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-1390
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Post-exercise Sport Students
Keywords: acupuncture; lactic acid levels; post-exercise recovery; press tack needle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Press tack needle acupuncture (Experimental)
  Interventions: Device: Press tack needle acupuncture
- Control (No Intervention)

INTERVENTIONS:
Device: Press tack needle acupuncture — Pyonex press tack needle sized 0.20x1.2mm
  Arms: Press tack needle acupuncture

SUMMARY:
Background: In sports, recovery after exercise is a very important process for athletes. Several studies have shown that the rate of disease associated with athlete's recovery can be increased by several modalities, one of which is acupuncture.

Objectives: The purpose of this study was to see how the effect of press tack needle acupuncture in reducing blood lactic acid levels after exercise in sports students.

Methods: The study design was a randomized controlled clinical trial. Twenty-four sport students were divided into two groups: the acupuncture group (n = 12) and the normal group (n = 12). Press tack needle was attached on PC6 Neiguan and ST36 Zusanli 30 minutes before doing high-intensity exercise. Measurement of lactic acid levels was carried out at 5 minutes and 30 minutes after exercise.

ELIGIBILITY:
Inclusion Criteria:

* willingness to fill out an informed consent form;
* age between 18-25 years;
* male;
* has a BMI value of 18.5-22.9 kg/m2;
* there is no history of injury or history of surgery on the lower extremities in the last three months;
* the individual is in good health.

Exclusion Criteria:

* absence or refusal to be examined and not cooperative.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Lactic acid levels | 5-minute after physical exercise and 30-minute after physical exercise
  Mean difference of lactic acid levels between two groups

SECONDARY OUTCOMES:
Heart rate | 0-minute after physical exercise and 30-minute after physical exercise
  Mean difference of heart rate between two group

CONTACTS AND LOCATIONS:
Locations (1):
- Fakultas Ilmu Keolahragaan Universitas Negeri Jakarta, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Djaali W, Mighra BA, Nurdin F, Setiakarnawijaya Y. Press-Tack Needle Acupuncture Reduces Postexercise Blood Lactic-Acid Levels in Sports Students. Med Acupunct. 2023 Oct 1;35(5):246-250. doi: 10.1089/acu.2023.0003. Epub 2023 Oct 17. PMID 37920859